CLINICAL TRIAL: NCT02706132
Title: MSC for ABO Incompatible Liver Transplantation
Brief Title: Therapeutic Strategy and the Role of Mesenchymal Stromal Cells for ABO Incompatible Liver Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yang Yang, Department of Liver Transplantation, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-08
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Liver Transplantation
Keywords: Mesenchymal stromal cells; Liver Transplantation; ABO blood group

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- The MSCs group (Experimental): The group of patients receive allogeneic MSCs therapies.
  Interventions: Biological: Mesenchymal Stem Cells(MSCs)

INTERVENTIONS:
Biological: Mesenchymal Stem Cells(MSCs) — Six doses of 1*10^6/kg body weight MSCs are given, intravenously.

SUMMARY:
The purpose of this study is to determine whether MSCs are safe and effective in reducing the primary nonfunction (PNF), acute rejection and Ischemic-type Biliary Lesions (ITBLs) morbidity in ABO-incompatible Liver Transplantation.

DETAILED DESCRIPTION:
ABO incompatible liver transplantations is considered to be a rescue option in emergency transplantation.The A、B antibodies to grafts bind to the graft endothelium and activate complement, which attracts and activates neutrophils and platelets and increases the permeability of the endothelium. The neutrophils exude, the platelets aggregate, and the small vessels of the graft get thrombosed, resulting in ischemic damage,leading nonfunction grafts.In addition, if the A、 B antibodies remain high level, it can lead to acute humoral immune rejection. A lot of research confirmed that the ABO incompatible is a risk factor of postoperative short- and long-term survival. And mesenchymal stromal cells (MSCs) are characterized by the properties of immunosuppressive and regenerative properties, which make MSCs great attractive in treating immunological diseases (including transplant rejection) and organ/tissue ischemic injury. So we conduct this clinical study,to confirm the effect of MSCs in ABO incompatible liver transplantation by comparing the incidence of primary nonfunction, acute rejection, biliary complications and survival rates.

ELIGIBILITY:
Inclusion Criteria:

* First liver transplantation with a ABO-incompatible graft(B→A，AB→A，A→B，AB→B，A→O，B→O，AB→O).
* Ages of 18 or older.
* Patients receive liver transplantation due to benign end stage liver disease.
* Patients or legal agent must be able to give informed consent.

Exclusion Criteria:

* Second or combined organ transplant recipient.
* Combined transplantations such as simultaneous liver/kidney transplants
* Malignant disease.
* Uncontrol bacterial, fungal, viral or parasitic infection.
* Withdraw or unable to finish the follow-up.
* Unwilling to sign informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy: one year graft survival rate | one year

SECONDARY OUTCOMES:
the rate of acute rejection | one year
the rate of ischemic-type biliary lesions | one year
safety: rate of (serious) adverse events in the study population | one year
  adverse events include: allergic reaction, prothrombotic effects, opportunistic infections and malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yang, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No